CLINICAL TRIAL: NCT02891941
Title: Neuroimaging & Plasma Markers for Predicting Outcomes After Mild Traumatic Brain Injury
Status: Terminated | Type: Observational
Why Stopped: Funding withdrawn
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00078556
Record Dates: First submitted 2013-09-19; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Traumatic Brain Injury; Injury of Body Region
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — whole blood, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mild Traumatic Brain Injury: This cohort will have sustained a closed head injury, defined as externally inflicted trauma without skull fracture within the last month.

SUMMARY:
This exploratory study aims to identify the most promising biomarkers that alone or in combination might predict development of mood disorders [i.e., major depression (MD], cognitive disorders [i.e., executive function deficits (EFD)], and functional impairment following repetitive/mild traumatic brain injury (MTBI).

DETAILED DESCRIPTION:
This will be a prospective study of subjects with MTBI, body injury and healthy controls. Subjects who meet the study criteria will be enrolled in the study after they provide informed consent.

All subjects will be followed longitudinally at 3 and 6 months post-injury.

All subjects will have 3-4 visits:

Screening visit to determine eligibility; first study visit within 1 month of injury for those with brain or body injury (at the time of screening or within 1 month of screening for healthy controls); second study visit at 3 months post-injury (3 months after the first visit for healthy controls) and third study visit at 6 months post-injury (6 months after the first visit for healthy controls).

ELIGIBILITY:
Inclusion Criteria:

Individuals with MTBI: Inclusion Criteria:

1. Have sustained a closed head injury, defined as externally inflicted trauma without skull fracture;
2. Have a Glasgow Coma Scale (GCS) score 13 or above
3. Meet the American Congress of Rehabilitation Medicine criteria for mild traumatic brain injury
4. Have experienced the last injury within 1 month
5. Be in excellent/good medical health as assessed by the General Medical Health Rating (GMHR) scale
6. Have sufficient cognitive capacity to provide informed consent
7. Be between 18-65 years of age and
8. Be willing to have brain MRI and a blood draw,

Individuals with Body Injury will meet inclusion criteria 4-8. Instead of criteria for head injury (1-3) they would have had body injury (defined as injury below the neck (e.g., limb fractures, stab wound abdomen).

Age, and sex, matched normal controls: Inclusion Criteria:

1. No history of head injury or any other types of brain injury
2. Inclusion criteria 5-8

Exclusion Criteria:

1. History of stroke, seizures or other pre-injury neurological diseases
2. Mental Retardation
3. History of skull fracture
4. Presence of severe unstable medical disease
5. Contraindications to the MRI brain scan
6. Possibility of pregnancy
7. Presence of communication difficulties, such as moderate to severe hearing or language impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency rooms, local physicians, free-standing urgent care establishments, local community
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Specific biomarkers (alone or in combination) assessed 3 months after MTBI | 3 months after MTBI.
  This exploratory study aims to identify the most promising biomarkers that alone or in combination might predict development of mood disorders [i.e., major depression (MD], cognitive disorders [i.e., executive function deficits (EFD)], and functional impairment following repetitive/MTBI. This will provide pilot data for a larger study with increased sample size and more stringent panel of markers based on results obtained.
Specific biomarkers (alone or in combination) assessed 6 months after MTBI. | 6 months after MTBI
  This exploratory study aims to identify the most promising biomarkers that alone or in combination might predict development of mood disorders [i.e., major depression (MD], cognitive disorders [i.e., executive function deficits (EFD)], and functional impairment following repetitive/MTBI. This will provide pilot data for a larger study with increased sample size and more stringent panel of markers based on results obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Vani Rao, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States